CLINICAL TRIAL: NCT04690023
Title: Comparison of Ultrasound-guided PENG Block and Supra-inguinal Fascia Iliaca Compartment Block for Postoperative Opioids Consumption and Early Motor Recovery After Total Hip Arthroplasty: a Randomized Controlled Non-inferiority Clinical Trial.
Brief Title: PENG Block vs Supra-inguinal Fascia Iliaca Compartment Block for Postoperative Opioids Consumption and Early Motor Recovery After THA: a Randomized Controlled Non-inferiority Clinical Trial.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Jean François Brichant, Head of Anesthesiology Departement, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2020/381
Record Dates: First submitted 2020-12-28; First posted 2020-12-30 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Total Hip Arthroplasty
MeSH Terms: interventions — Dental Occlusion

STUDY DESIGN:
Intervention Model Description: Non-inferiority randomized controlled clinical trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Non-inferiority controlled RCT with two groups simple-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENG block (Active Comparator): Patients scheduled for total hip arthroplasty with spinal anesthesia receive before intra-thecal injection, ultrasound-guided PENG block. Patients in PENG group receive multimodal postoperative analgesia techniques coupled with morphine PCA pump.
  Interventions: Procedure: Pericapsular nerves group (PENG) block; Drug: Ropivacaine 0,75% in PENG block
- SFICB block (Active Comparator): Patients scheduled for total hip arthroplasty with spinal anesthesia receive before intra-thecal injection, ultrasound-guided supra-inguinal fascia iliaca compartment block. Patients in SFICB group receive multimodal postoperative analgesia techniques coupled with morphine PCA pump.
  Interventions: Procedure: Supra-inguinal fascia-iliaca compartment block; Drug: Ropivacaine 0,375% in SFICB block

INTERVENTIONS:
Procedure: Pericapsular nerves group (PENG) block — Patients scheduled for total hip arthroplasty with spinal anesthesia receive before intra-thecal injection, ultrasound-guided PENG block with injection 20 ml of ropivacaine 0,75%, between the anterior hip articular capsule, the ilii-psoas muscle, the ileo-pubic eminence and the antero-inferior iliac spine.
  Arms: PENG block
Procedure: Supra-inguinal fascia-iliaca compartment block — Patients scheduled for total hip arthroplasty with spinal anesthesia receive before intra-thecal injection, ultrasound-guided supra-inguinal fascia iliaca compartment block with injection over de inguinal ligament of 40 ml of ropivacaine 0,375%, between de ilio-psoas muscle and internal oblique muscle.
  Arms: SFICB block
Drug: Ropivacaine 0,75% in PENG block — 20 ml injection of ropivacaine 0,75%
  Arms: PENG block
Drug: Ropivacaine 0,375% in SFICB block — 40 ml injection of ropivacaine 0,375%
  Arms: SFICB block

SUMMARY:
To compare the impact of pericapsular nerve group block (PENG) versus the supra-inguinal fascia-iliaca compartment block (SFICB) in postoperative analgesia, opioid sparing and enhanced recovery after surgery of total hip arthroplasty by poster-lateral approach.

DETAILED DESCRIPTION:
ASA physical status 1, 2 and 3 patients scheduled to undergo elective total hip arthroplasty by poster-lateral (Moore) surgical approach with spinal anesthesia.

The investigators want to confirm the non-inferiority of the SFICB compared to the PENG block on postoperative first 6 hours after surgery NRS pain score and 48 hours opioids consumption, and the difference between these in terms of early recovery and motor impact on two first day after surgery. The principal investigator perform these regional anesthesia techniques with ultrasound guided injections.

ELIGIBILITY:
Inclusion Criteria:

- Adults patients scheduled to undergo elective primary total hip arthroplasty by posterior surgical approach with spinal anesthesia

Exclusion Criteria:

* Patient refusal
* Allergy to administrated drugs or local infection
* Pregnancy
* History of chronic pain
* Drugs addiction
* Mental ou neurological diseases
* Kidney or liver serious diseases

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
NRS 6 hours | 6 hours after surgery
  The primary endpoint of the study will be the between-group comparisons in postoperative NRS pain scores on 0 to 10 scale.

SECONDARY OUTCOMES:
6 minutes walk test | 48 jours after surgery
  Difference in traveled distance (metres) at six minutes walking test 48 hours after surgery
Opioids secondaires side effects | 48 hours after surgery
  Incidence of morphine related side effects in two groups
QoR-15 | 72 hours after surgery
  QoR-15 French validated questionnaire for the evaluation of recovery after surgery
2 minutes walk test | 24 hours after surgery
  Difference in traveled distance (metres) at two minutes walking test 24 hours after surgery
Opioid sparing | 48 hours after intervention
  Difference in cumulated morphine consumption in first 48 hours after surgery
DN4 | 72 hours after surgery
  Difference between the two groups in the DN4 questionnaire to assess the risk of persistent pain after surgery.
IPO | 72 hours after surgery
  Pain management satisfaction score by revised American Pain Society Patient Outcomes Questionnaire (APS- POQ-R).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657
- [Background] Vermeylen K, Desmet M, Leunen I, Soetens F, Neyrinck A, Carens D, Caerts B, Seynaeve P, Hadzic A, Van de Velde M. Supra-inguinal injection for fascia iliaca compartment block results in more consistent spread towards the lumbar plexus than an infra-inguinal injection: a volunteer study. Reg Anesth Pain Med. 2019 Feb 22:rapm-2018-100092. doi: 10.1136/rapm-2018-100092. Online ahead of print. PMID 30798268